CLINICAL TRIAL: NCT05936489
Title: A Prospective, Single-Center, Open-Label, Study of the Plasma Pharmacokinetics and Safety Following Topical Administration of LNZ101 and LNZ100 Ophthalmic Solutions in Healthy Adult Subjects With Presbyopia
Brief Title: Plasma Pharmacokinetics and Safety of LNZ101 and LNZ100 Ophthalmic Solutions in Healthy Adult Subjects With Presbyopia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LENZ Therapeutics, Inc (Other)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-100-0007
Record Dates: First submitted 2023-06-21; First posted 2023-07-07 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Eye Diseases; Presbyopia; Refractive Errors; Brimonidine Tartrate; Aceclidine; Ophthalmic Solutions
MeSH Terms: conditions — Eye Diseases; Presbyopia; Refractive Errors | interventions — aceclidine; Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: A Prospective, Single-Center, Open-Label, Study of the Plasma Pharmacokinetics
Masking Description: this is an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LNZ101 (Other): Aceclidine 1.75% / Brimonidine combination (non-preserved) ophthalmic solution
  Interventions: Drug: Aceclidine + Brimonidine
- LNZ100 (Other): Aceclidine 1.75% (non-preserved) ophthalmic solution
  Interventions: Drug: Aceclidine

INTERVENTIONS:
Drug: Aceclidine + Brimonidine — LNZ101 (Aceclidine/Brimonidine) non-preserved ophthalmic solution
  Arms: LNZ101
Drug: Aceclidine — LNZ100 (Aceclidine) non-preserved ophthalmic solution
  Arms: LNZ100

SUMMARY:
This is a single-center, open-label, randomized study to assess the plasma pharmacokinetic profile of LNZ101 and LNZ100.

DETAILED DESCRIPTION:
To characterize the plasma pharmacokinetics and safety profile of LNZ101 and LNZ100 ophthalmic solutions in both eyes once a day for 8 days in healthy volunteers with presbyopia

ELIGIBILITY:
Inclusion Criteria:

* Each subject must:

  1. Be able and willing to provide written informed consent and sign a Health Information Portability and Accountability Act (HIPAA) form prior to any study procedure being performed;
  2. Be able and willing to follow all instructions and attend all study visits;
  3. Be 45-75 years of age of either sex and any race or ethnicity;
  4. Be presbyopic in both eyes;

Exclusion Criteria:

* Each subject must not:

  1. Have known contraindications or sensitivity to the use of the investigational drug or its components, or any other medications required by the protocol;
  2. Have any active systemic or ocular disorder other than refractive disorder;
  3. Have prior, current or anticipated use of any contact lenses during study participation;
  4. Have presence of any abnormality of the lids, ocular surface, or lacrimal duct system that could affect ophthalmic drop absorption;
  5. Have anticipated inability to stay confined on required study days;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 and Day 8
  Maximum plasma concentrations of LNZ100 and LNZ101
Tmax | Day 1 and Day 8
  Time of maximum plasma concentrations of LNZ100 and LNZ101
AUC0-t | Day 1 and Day 8
  Area under the concentration-time curve from time 0 to time t of LNZ100 and LNZ100
AUC0-inf | Day 1 and Day 8
  Area under the concentration-time curve from time 0 to infinity of LNZ100 and LNZ101
T1/2 | Day 1 and Day 8
  Terminal half-life of LNZ100 and LNZ101

OTHER OUTCOMES:
Safety: adverse event reporting | up to 37 days
  The number of patients who experience one or more TEAE during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Kris Gameblin, Study Director — LENZ Therapeutics
Locations (1):
- Site #101, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan.